CLINICAL TRIAL: NCT05262764
Title: Post Marketing Surveillance on Long Term Drug Use of JARDIANCE® Tablets in Patients With Chronic Heart Failure in Japan
Brief Title: Post Marketing Surveillance (PMS) of JARDIANCE in Chronic Heart Failure (CHF)
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0286
Record Dates: First submitted 2022-03-01; First posted 2022-03-02 (Actual); Results first posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — empagliflozin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- JARDIANCE®: Patients in Japan with chronic heart failure who were prescribed JARDIANCE® tablets and who were never treated with Empagliflozin before enrolment. Treatment was in accordance with the latest guidelines from The Japanese Circulation Society (JCS). Patients were observed for up to 52 weeks after start of the treatment or until discontinuation of administration.
  Interventions: Drug: JARDIANCE®

INTERVENTIONS:
Drug: JARDIANCE® — Treatment was in accordance with the latest guidelines from The Japanese Circulation Society (JCS).
  Other Names: empagliflozin

SUMMARY:
Study objective is to investigate the safety and effectiveness of long-term daily use of JARDIANCE® Tablets in patients with chronic heart failure (CHF) under real-world use.

ELIGIBILITY:
Inclusion Criteria:

* Patients with chronic heart failure (CHF) failure who are prescribed with JARDIANCE® Tablets in Japan
* Patients who have never been treated with Empagliflozin (including treatment for type 2 diabetes mellitus (T2DM)) before enrolment

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients with chronic heart failure (CHF).
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-06-28 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nippon Boehringer Ingelheim Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
Once the criteria in section "Time Frame" are fulfilled, researchers can use the following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement". Furthermore, researchers can request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After structured results have been posted, all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents -upon signing of a 'Document Sharing Agreement'.For study data -1. after the submission and approval of the research proposal (checks will be performed by the sponsor and/or the independent review panel, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a legal agreement.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] Yamamoto K, Naito Y, Watanabe S. Safety and effectiveness of empagliflozin in Japanese patients with heart failure: a 1-year post-marketing surveillance study stratified by age. Expert Opin Drug Saf. 2025 Jun 18:1-9. doi: 10.1080/14740338.2025.2519835. Online ahead of print. PMID 40512403
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Pre-assignment Details: This was a non-interventional, single arm study based on newly collected data Patients were observed for up to 52 weeks after start of the treatment with JARDIANCE® Tablets or until discontinuation of administration.
Groups:
- JARDIANCE®: Patients in Japan with chronic heart failure who were prescribed JARDIANCE® (Empagliflozin) tablets and who were never treated with Empagliflozin before enrolment (including treatment for type 2 diabetes mellitus). Treatment was in accordance with the latest guidelines from The Japanese Circulation Society (JCS). Patients were observed for up to 52 weeks after start of the treatment or until discontinuation of administration.
Period: Overall Study
Arm/Group | JARDIANCE®
Started (Registered participants) | 1200
Safety Set | 1166
Completed (Participants in effectiveness set) | 1165
Not Completed | 35
Not completed — Case report form not collected | 9
Not completed — No patient visits after entry | 23
Not completed — Registration rule not followed | 2
Not completed — Patient of non-chronic heart failure | 1

BASELINE CHARACTERISTICS:
Population: Safety set: all patients who didn't have important Protocol Deviations regarding safety and regulatory issues.
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 1166
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.9 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 455
  Male | 711
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Adverse Drug Reactions (ADRs)
Description: Number of subjects with ADRs (focus on hypoglycaemia, the events relevant for volume depletion, influence of ketone body increased / ketoacidosis, renal impairment).
Time Frame: Up to 52 weeks
Population: Safety set: all patients who didn't have important Protocol Deviations regarding safety and regulatory issues.
Measure: Count of Participants; unit: Participants
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 1166
Participants | 61

2. Secondary Outcome: Incidence of All-cause Death
Description: Incidence of all-cause death.
Time Frame: Up to 52 weeks
Population: Safety set: all patients who didn't have important Protocol Deviations regarding safety and regulatory issues.
Measure: Number (95% Confidence Interval); unit: Deaths per 100 person-years
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 1166
Deaths per 100 person-years | 3.01 [2.03 to 4.29]

3. Secondary Outcome: Incidence of Cardiovascular Death
Description: Incidence of cardiovascular death.
Time Frame: Up to 52 weeks
Population: Safety set: all patients who didn't have important Protocol Deviations regarding safety and regulatory issues.
Measure: Number (95% Confidence Interval); unit: Deaths per 100 person-years
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 1166
Deaths per 100 person-years | 0.90 [0.41 to 1.71]

4. Secondary Outcome: Incidence of Hospitalizations for Heart Failure
Description: Incidence of hospitalizations for heart failure.
Time Frame: Up to 52 weeks
Population: Safety set: all patients who didn't have important Protocol Deviations regarding safety and regulatory issues.
Measure: Number (95% Confidence Interval); unit: 1st Hospitalization per 100 person-years
Arm/Group | JARDIANCE®
Number analyzed (Participants) | 1166
1st Hospitalization per 100 person-years | 2.53 [1.64 to 3.74]

ADVERSE EVENTS:
Time Frame: Up to 52 weeks.
Description: Safety set: All patients who didn't have important Protocol Deviations regarding safety and regulatory issues.
Arm/Group | JARDIANCE®
All-Cause Mortality (participants affected / at risk) | 30/1166
Serious Adverse Events (participants affected / at risk) | 148/1166
Other Adverse Events (participants affected / at risk) | 0/1166
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JARDIANCE® (N=1166)
Anaemia (Blood and lymphatic system disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 2
Aortic valve incompetence (Cardiac disorders) | 1
Arrhythmia (Cardiac disorders) | 1
Atrial fibrillation (Cardiac disorders) | 7
Bradycardia (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 2
Cardiac failure (Cardiac disorders) | 58
Cardiac failure acute (Cardiac disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 5
Cardiac failure congestive (Cardiac disorders) | 3
Cardiac sarcoidosis (Cardiac disorders) | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 1
Cardio-respiratory arrest (Cardiac disorders) | 2
Cardiomyopathy (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Sinus node dysfunction (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Enterocolitis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Inguinal hernia (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 1
Large intestine perforation (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Cardiac death (General disorders) | 1
Death (General disorders) | 2
Prosthetic cardiac valve thrombosis (General disorders) | 1
Sudden cardiac death (General disorders) | 1
Sudden death (General disorders) | 2
Bile duct stone (Hepatobiliary disorders) | 2
Cholangitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Abdominal wall abscess (Infections and infestations) | 1
Abscess (Infections and infestations) | 1
Arthritis bacterial (Infections and infestations) | 1
COVID-19 (Infections and infestations) | 6
Escherichia bacteraemia (Infections and infestations) | 1
Liver abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 6
Pneumonia aspiration (Infections and infestations) | 4
Pneumonia bacterial (Infections and infestations) | 1
Psoas abscess (Infections and infestations) | 1
Pyelonephritis (Infections and infestations) | 2
Pyelonephritis acute (Infections and infestations) | 1
Sepsis (Infections and infestations) | 3
Septic shock (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 2
Femoral neck fracture (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Near drowning (Injury, poisoning and procedural complications) | 1
Radius fracture (Injury, poisoning and procedural complications) | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1
Blood pressure decreased (Investigations) | 1
Blood urea increased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 2
Dehydration (Metabolism and nutrition disorders) | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 1
Marasmus (Metabolism and nutrition disorders) | 1
Immobilisation syndrome (Musculoskeletal and connective tissue disorders) | 1
Angioimmunoblastic T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Cerebellar haemorrhage (Nervous system disorders) | 2
Cerebral infarction (Nervous system disorders) | 6
Depressed level of consciousness (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 1
Embolic cerebral infarction (Nervous system disorders) | 1
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 2
Subarachnoid haemorrhage (Nervous system disorders) | 2
Taste disorder (Nervous system disorders) | 1
Thrombotic cerebral infarction (Nervous system disorders) | 1
Delirium (Psychiatric disorders) | 1
Transient psychosis (Psychiatric disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 4
Azotaemia (Renal and urinary disorders) | 1
Chronic kidney disease (Renal and urinary disorders) | 2
Renal disorder (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
Aortic dissection (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1

LIMITATIONS AND CAVEATS:
Since this surveillance was an observational, non-interventional study, it lacked the methodological rigour of a randomised controlled trial. The study was conducted in an unblinded manner and without controls.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2024-04-01): https://cdn.clinicaltrials.gov/large-docs/64/NCT05262764/Prot_000.pdf
  • Statistical Analysis Plan (2024-08-14): https://cdn.clinicaltrials.gov/large-docs/64/NCT05262764/SAP_001.pdf